CLINICAL TRIAL: NCT02586090
Title: Innovative Approaches to Adolescent Obesity Treatment: Exploring the Role of Parents
Brief Title: The Role of Parents in Adolescent Obesity Treatment
Acronym: TEENS+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20005235; 1R21HD084930 (NIH)
Record Dates: First submitted 2015-07-16; First posted 2015-10-26 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Pediatric Obesity
Keywords: Pediatric Obesity; Lifestyle Intervention; Family-based Intervention; Motivational Interviewing
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Assessors blind to hypotheses and allocation Interventionsts blinded to hypotheses
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parents as Coaches (Active Comparator): PAC (modeled after NIH-funded NOURISH) focuses on parenting strategies to support and facilitate their child's weight management via family-based change. Each visit includes group psychoeducation and discussion, focused on parenting strategies to facilitate healthy weight management in their child(ren). Topics include focus such as role modeling, strategies for healthy lifestyle changes, and how to be a coach to your teen.
  Interventions: Behavioral: Parents as Coaches
- Parent Weight Loss (Experimental): In PWL parents will be given a weight loss goal of 1-2 lbs/week, as well as specific calorie and fat prescriptions, PA goals, and instructions to self-monitor key information. Parents will receive training in core behavioral weight loss strategies (e.g., goal setting, stimulus control) and techniques to help them achieve these goals and will also receive personalized feedback throughout the program
  Interventions: Behavioral: Parent Weight Loss

INTERVENTIONS:
Behavioral: Parents as Coaches — PAC (modeled after NIH-funded NOURISH) focuses on parenting strategies to support and facilitate their child's weight management via family-based change. Each visit includes group psychoeducation and discussion, focused on parenting strategies to facilitate healthy weight management in their child(ren). Topics include focus such as role modeling, strategies for healthy lifestyle changes, and how to be a coach to your teen.
  Arms: Parents as Coaches
Behavioral: Parent Weight Loss — In PWL parents will be given a weight loss goal of 1-2 lbs/week, as well as specific calorie and fat prescriptions, PA goals, and instructions to self-monitor key information. Parents will receive training in core behavioral weight loss strategies (e.g., goal setting, stimulus control) and techniques to help them achieve these goals and will also receive personalized feedback throughout the program
  Arms: Parent Weight Loss

SUMMARY:
The study will pilot a randomized control trial to investigate the feasibility and preliminary efficacy of two distinct parent treatments on a dietary intervention for overweight and obese adolescents.

DETAILED DESCRIPTION:
Investigators will recruit overweight or obese adolescents (BMI >85th percentile) and parent(s) (BMI >25 kg/m2). Families will participate in one of two 4-month treatments: 1) TEENS+Parents as Coaches (PAC), engaging parents as helpers in their child's weight management, or 2) TEENS+Parent Weight Loss (PWL), engaging parents in their own weight management. All adolescents will participate in TEENS+, which includes behavioral support, nutrition education, and supervised physical activity.

For the adolescents, intervention will consist of weekly 1 hour exercise sessions and alternating weekly 1 hour behavioral and nutrition group sessions. Parents will also attend the nutrition sessions and participate in a behavioral parent-only biweekly group. Parent behavioral group sessions will be specific to the treatment arm (e.g. PAC or PWL). Assessments will consist of anthropometric measures, psychological surveys, and nutritional evaluations. Assessments will be completed at baseline, post-test and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Adolescent Inclusion Criteria:

* BMI ≥85% percentile for age and gender according to the CDC Growth Charts
* Age 12 to 16
* must reside with the primary participating parent
* parent must have a BMI ≥25 kg/m 2
* parent must be willing to participate in the protocol

Parent Inclusion Criteria:

* 18-60 years of age
* BMI ≥25 kg/m2
* must reside with the adolescent

Exclusion Criteria:

Adolescent Exclusion Criteria

* non-English speaking
* medical condition(s) that may be associated with unintentional weight change
* use of oral glucocorticoids, atypical antipsychotics, weight loss medications, or an investigational medication within 3 months of study participation;
* medical condition(s) that may be negatively impacted by exercise
* psychiatric, cognitive, physical or developmental conditions that would impair the ability to complete assessments, participate in a group, or conduct physical activity
* reports of compensatory behaviors in the past 3 months
* current pregnancy or plan to become pregnant during study period
* previous participation in HM11113, HM13833, HM20003076, IRB3008, IRB6255, HM11390, HM13468, HM14973 or HM14139
* current participation in another weight loss program; or 11) personal history of weight loss surgery.
* clinically significant depression
* clinically significant eating disorder
* change in dose of metformin, oral contraceptives, tricyclic antidepressants (TCAs), selective serotonin reuptake inhibitors (SSRIs), or stimulant medications within 3 months prior to study participation.
* weight in excess of 400 pounds
* admission to a psychiatric hospital within the past year

Parent Exclusion Criteria

* non-English speaking
* medical condition(s) that may be associated with unintentional weight change
* use of oral glucocorticoids, atypical antipsychotics, weight loss medications, or investigational medications within 3 months of study participation
* psychiatric, cognitive, physical or developmental conditions that would impair the parent's ability to respond to assessments, participate in physical activity or participate in a group
* reports of compensatory behaviors in the past 3 months
* current pregnancy, lactation, less than 6 months post-partum, or plan to become pregnant during the study period
* past participation in IRB3354, HM11113, HM13833, HM20003076, IRB3008, IRB6255, HM11390, HM13468, HM14973 or HM14139
* currently engaged in another weight loss program, or 9) personal history of weight loss surgery.
* Severe depression or endorsing suicidal thoughts
* admission to a psychiatric hospital within the past year.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Between-group differences in parent weight change. | 4 months (pre-intervention - post-test)
  Weight change (kg; parents)- primary outcome; trial is powered on parent weight change
Within group differences in adolescent changes in BMI | 4 months (pre-intervention - post-test)
  BMI change (kg/m2; adolescent)

SECONDARY OUTCOMES:
Changes in parent dietary intake | 4 months (pre-intervention - post-test)
  Average total energy intake (kcal/day) estimated via 3-day food record
Changes in authoritative parenting (API) and parent feeding practices measured via Child Feeding Questionnaire | 4 months (pre-intervention - post-test)
  parenting and feeding style
Changes in child dietary intake | 4 months (pre-intervention - post-test)
  Average total energy intake (kcal/day) estimated via 3-day food record
Changes in parent physical activity | 4 months (pre-intervention - post-test)
  Mean total daily energy expenditure (kcal/day) estimated via accelerometer
Changes in adolescent physical activity | 4 months (pre-intervention - post-test)
  Mean total daily energy expenditure (kcal/day) estimated via accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Bean, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU Healthy Lifestyles Center, Henrico, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form: Consent Form (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02586090/ICF_002.pdf
  • Informed Consent Form: Assent Form (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02586090/ICF_003.pdf